CLINICAL TRIAL: NCT03854253
Title: Effect of Introducer Length on the Rate of Radial Artery Occlusion During Endovascular Coronary Procedures: а Pilot Randomized Clinical Trial
Brief Title: Effect of Introducer Length on the Rate of Radial Artery Occlusion During Endovascular Coronary Procedures
Acronym: IntroLength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IntroLength
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long introducer 6Fr-25cm (Experimental): The investigators will perform transradial coronary angiography and percutaneous coronary interventions using long introducer sheath 6Fr-25cm
  Interventions: Procedure: Long introducer sheath
- Short introducer 6Fr-10cm (Active Comparator): The investigators will perform transradial coronary angiography and percutaneous coronary interventions using short introducer sheath 6Fr-10cm
  Interventions: Procedure: Short introducer sheath

INTERVENTIONS:
Procedure: Long introducer sheath — The investigators will perform transradial coronary angiography and percutaneous coronary interventions using introducer sheath 6Fr-25cm
  Arms: Long introducer 6Fr-25cm
Procedure: Short introducer sheath — The investigators will perform transradial coronary angiography and percutaneous coronary interventions using introducer sheath 6Fr-10cm
  Arms: Short introducer 6Fr-10cm

SUMMARY:
This study evaluates estimate impact of introducers length during endovascular coronary procedures on rate of a radial artery occlusion. For half of participants will use short introducers, while for other will use long introducers during transradial coronary intervention.

DETAILED DESCRIPTION:
The transradial approach for coronary angiography and interventions is increasingly utilized around the world. Radial artery occlusion is the most common significant complication after transradial catheterization, with incidence varying between 1% and 10%. Endothelial injury of the radial artery and decrease in blood flow after sheath and catheter insertion appear to contribute to thrombus formation and are predisposing factors for radial artery occlusion. Procedural factors can predict and influence radial artery occlusion incidence. Sheath size and its relation to radial artery diameter, as well as the utilization of specific pharmacological agents (such as anticoagulants and vasodilators) have been studied. But, impact of Introducer sheath length on the rate of a radial artery occlusion has not been studied. The investigators suggest that, longer introducer sheath sizes can prevented the vascular damage and a pro-thrombotic environment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Applicability of transradial approach

Exclusion Criteria:

* Failure of the transradial approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Popov, Principal Investigator — Tomsk National Research Medical Center of the Russian Academy of Sciences
Locations (1):
- Tyumen Cardiology Research Center, Tomsk National Research Medical Center, Russian Academy of Science, Tyumen, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Started | 50 | 50
Completed | 49 | 50
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: One hundred patients who underwent coronary angiography (CAG) and/or percutaneous coronary intervention (PCI) with a transradial approach at the Cardiology Research Center in 2019 were enrolled in the study and randomized into two groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 30 | 67
  >=65 years | 13 | 20 | 33
Age, Continuous [Median (Standard Deviation); unit: years] | 58.04 (11.163) | 63.46 (9.265) | 60.75 (10.563)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 35 | 28 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 50 | 50 | 100
Region of Enrollment [Number; unit: participants]
  Russia | 50 | 50 | 100
Signed informed consent document [Count of Participants; unit: Participants] | 50 | 50 | 100
Repeated radial access [Count of Participants; unit: Participants] | 14 | 19 | 33
Diabetes mellitus [Count of Participants; unit: Participants] | 11 | 10 | 21
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (5.5) | 31.8 (6.2) | 31.6 (5.8)
Taking anticoagulants [Count of Participants; unit: Participants] — Participants who took anticoagulants
  Participants | 11 | 19 | 30
CAG [Count of Participants; unit: Participants] — Patients who underwent coronary angiography (CAG) .
  Participants | 44 | 39 | 83
PCI [Count of Participants; unit: Participants] — Participants who underwent percutaneous coronary intervention (PCI).
  Participants | 4 | 5 | 9
Ad hoc PCI [Count of Participants; unit: Participants] — Participants who underwent immediate PCI after CAG.
  Participants | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radial Artery Occlusion
Description: Participants who diagnosed a radial artery occlusion with color Doppler ultrasound.
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
Participants | 4 | 2

2. Secondary Outcome: Number of Participants With a Hematoma, Stage I
Description: Rate of access site complications during percutaneous procedures performed via a transradial approach. Local hematomas are classified according to the following scale: I - diameter not more than 5 cm, II - not more than 10 cm, III - not more than 10 cm, but not higher than the elbow, IV - above the elbow, V - with the threat of hand ischemia [Bertrand, O. F., De Larochelliere, R., Rodes-Cabau, J., Proulx, G., Gleeton, O., Manh Nguyen, C., Dery J.P., Barbeau G., Noel B., Larose E., Poirier P., Roy L. A Randomized Study Comparing Same-Day Home Discharge and Abciximab Bolus Only to Overnight Hospitalization and Abciximab Bolus and Infusion After Transradial Coronary Stent Implantation. Circulation, 2006 114(24), 2636-2643.doi:10.1161/circulationaha.106.638627]. Hematomas more than stage I were not recorded in both groups.
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
Participants | 8 | 8

3. Secondary Outcome: Rate of Conversion of Needle Type
Description: Rate of conversion type of Needle type during percutaneous procedures performed via a transradial approach.
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
Participants | 5 | 0

4. Secondary Outcome: Time of the Introducer Insertion
Description: Time from start punction of the radial artery to full insertion of the introducer
Time Frame: up to 10 days
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
seconds | 94 [67.5 to 162.5] | 42.5 [33 to 65.3]

5. Secondary Outcome: Time of the Procedure
Description: Time from insertion of the introducer to finish the procedure
Time Frame: up to 10 days
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
seconds | 448 [337.5 to 633] | 350.5 [307 to 506.8]

6. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy time, sec
Time Frame: up to 10 days
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
seconds | 82.0 [48.5 to 133.0] | 69.5 [48.0 to 118.3]

7. Secondary Outcome: Total Air Kerma
Description: Total air kerma, mGy
Time Frame: up to 10 days
Measure: Median (Standard Deviation); unit: mGy
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
mGy | 140.8 (97.7) | 128.2 (71.3)

8. Secondary Outcome: Number of Participants With a Perforation / Dissection of a Radial Artery.
Description: Rate of access site complications during percutaneous procedures performed via a transradial approach
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Median Nerve Neuritis
Description: Rate of access site complications during percutaneous procedures performed via a transradial approach
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With a Bleeding of the Puncture Site.
Description: Rate of access site complications during percutaneous procedures performed via a transradial approach.
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
Number analyzed (Participants) | 49 | 50
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected is 10 days.
Arm/Group | Long Introducer 6Fr-25cm | Short Introducer 6Fr-10cm
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50

LIMITATIONS AND CAVEATS:
For the analysis of results in the main group, 1 participant was unavailable due to transfer to another hospital because of developed acute cerebrovascular accident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03854253/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03854253/SAP_001.pdf